CLINICAL TRIAL: NCT03798847
Title: Safety and Performance of Journey II XR Total Knee System. A Retrospective, Multicenter Study
Brief Title: Safety and Performance of Journey II XR Total Knee System
Acronym: JIIXR
Status: Completed | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: JIIXR.PMCF.2018.13
Record Dates: First submitted 2018-11-27; First posted 2019-01-10 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Journey II XR Total Knee System
Keywords: Journey II XR Total Knee System

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Journey II XR TKA — Journey II XR Total Knee System

SUMMARY:
The objective of this study is to estimate the safety and performance of Journey II XR TKS based on retrospective data.

ELIGIBILITY:
Inclusion Criteria:

* Subject received primary uni- or bi-lateral total knee arthroplasty with the Journey II XR TKS for approved indication;
* The TKA occurred at least 12 weeks prior to enrollment.

Exclusion Criteria:

- None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subject received primary uni- or bi-lateral total knee arthroplasty with the Journey II XR TKS for approved indication
Sampling Method: Non-Probability Sample
Enrollment: 683 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Revision of one or more study device components | 12 weeks follow up
  Measure of the number of revision cases

SECONDARY OUTCOMES:
Adverse Events | 12 weeks follow up
  All collected and reported AEs
Health care utilization: Hospitalization | implantation through study completion, approximately 3 years
  Length of hospital stay for primary (index) surgery
Health care utilization: Hospitalization | Implantation through study completion, approximately 3 years
  Hospitalizations (admission for inpatient care) occurring after the hospitalization for the index surgery (number and length of stay)
Health care utilization: Rehabilitation | Implantation through study completion, approximately 3 years
  number of sessions and duration of rehabilitation in weeks
Health care utilization: Outpatient visits | Implantation through study completion, approximately 3 years
  Number and type of outpatient visits
Health Care Utilization: Re-operations | Implantation through study completion, approximately 3 years
  Number of re-operations and revisions
Quality of Life: EQ-5D-3L | Implantation through study completion, approximately 3 years
  EuroQol Five Dimensions Questionnaire
Quality of Life: KSS | Implantation through study completion, approximately 3 years
  2011 Knee Society Score
Return to Work | Implantation through study completion, approximately 3 years
  Changes in employment status will be recorded with the date on which the change occurred and the change status.
Technical Difficulties Encountered During Device Implantation | Implantation through study completion, approximately 3 years
  Number of technical difficulties encountered with the device

CONTACTS AND LOCATIONS:
Locations (12):
- United States (12):
  - Orthopedic Institute of the West, Phoenix, Arizona
  - Rush Copley Orthopaedics, Aurora, Illinois
  - Jerry Orthopaedic Institute, Port Huron, Michigan
  - Reno Orthopedic Clinic, Reno, Nevada
  - Orthopaedic Center of New Jersey, Somerset, New Jersey
  - Hospital for Joint Diseases Orthopaedics Institute, New York, New York
  - Regenerative Orthopedic Center (ROC), Oregon City, Oregon
  - Oregon Health & Science University, Portland, Oregon
  - San Antonio Orthopaedic Specialists, San Antonio, Texas
  - Anderson Orthopaedic Clinic, Alexandria, Virginia
  - Scott Orthopedic Center, Huntington, West Virginia
  - Aurora Medical Center, Kenosha, Wisconsin

IPD SHARING:
Plan to Share IPD: No